CLINICAL TRIAL: NCT01591135
Title: A Phase III Randomized Clinical Trial of Comparing Paclitaxel Plus 5-Fluorouracil Versus Cisplatin Plus 5-Fluorouracil in Chemoradiotherapy for Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Phase III Study of Comparing Paclitaxel Plus 5-Fluorouracil Versus Cisplatin Plus 5-Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Xiamen University (Other); Fujian Cancer Hospital (Other Government); Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai1
Record Dates: First submitted 2012-04-18; First posted 2012-05-03 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; chemoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Fluorouracil; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin (Active Comparator): Chemoradiotherapy with cisplatin and 5-fluorouracil for 2 cycles followed by adjuvant chemotherapy for 2 cycles.
  Interventions: Drug: Cisplatin plus 5-fluorouracil; Radiation: Radiation therapy
- Paclitaxel (Experimental): Patients randomized in Arm B will receive chemoradiation with weekly paclitaxel and 5-fluorouracil for 5 weeks followed by adjuvant chemotherapy with paclitaxel and 5-fluorouracil for 2 cycles.
  Interventions: Drug: Paclitaxel plus 5-fluorouracil; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Paclitaxel plus 5-fluorouracil — 5-ﬂuorouracil 300 mg/m2, d1-4, continuous infusion for 96 hours and paclitaxel 50 mg/m2 over 3 hours, d1 (week 1, week 2, week 3, week 4 and week 5); 5-ﬂuorouracil 600 mg/m2/d d1-3 and paclitaxel 175 mg/m2 d1(week 9 and week 13).
  Arms: Paclitaxel
Drug: Cisplatin plus 5-fluorouracil — cisplatin 25 mg/m2/d, d1-3, once every 4 weeks for 4 cycles (week 1, week 5, week 9 and week 13); 5-FU 600 mg/m2/d, d1-3, continuously infusion for 72 hrs,once every 4 weeks for 4 cycles (week 1, week 5, week 9 and week 13).
  Arms: Cisplatin
Radiation: Radiation therapy — A total dose of 61.2 Gy will be delivered in 34 fractions at 1.8 Gy/fraction, 5 fractions per week in 6.8 weeks.
  Arms: Cisplatin
Radiation: Radiation therapy — A total dose of 61.2 Gy will be delivered in 34 fractions at 1.8 Gy/fraction, 5 fractions per week in 6.8 weeks.
  Arms: Paclitaxel

SUMMARY:
The primary objective of this trial is to study whether paclitaxel plus 5-fluorouracil has better overall survival than cisplatin plus 5-fluorouracil in chemoradiotherapy for patients with locally advanced esophageal squamous cell carcinoma. 436 patients will be recruited into this study.

DETAILED DESCRIPTION:
Locally advanced esophageal squamous cell carcinoma. T2-4N0-1M0-1a,TxN1M0-1a，TxNxM1a （according to AJCC2002）

Scheme:

Eligible recurrent patients with esophageal cancer will first be stratified by nodal staging (N0 or N1), then randomized to 2 arms at 1:1 ratio.

Arm Cisplatin:

Chemoradiotherapy with cisplatin and 5-fluorouracil for 4 cycles.

Arm Paclitaxel:

Chemoradiotherapy with weekly paclitaxel and 5-fluorouracil for 5 weeks followed by adjuvant chemotherapy for 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age 18-75
* Both genders
* Esophageal squamous cell carcinoma confirmed by pathology
* Local advanced esophageal squamous cell carcinoma (T2N0M0-TxNxM1a, AJCC 2002)
* No radiotherapy, chemotherapy or other treatments prior to enrollment
* PS ECOG 0-2
* Life expectancy of more than 3 months
* Hemoglobin（Hb）≥9 g/dL
* WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L
* platelet count (Pt) ≥100x 109/L
* Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL<1.5 x ULN
* Renal function: creatinine < 1.5 x ULN
* No immuno-deficiency
* Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

* Complete esophageal obstruction
* Deep esophageal ulcer
* Esophageal perforation
* Haematemesis
* After surgery, exploratory thoracotomy, radiotherapy, chemotherapy, or targeting therapy
* Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years
* Participation in other interventional clinical trials within 30 days
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Drug addiction
* Alcoholism or AIDS
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* Patient who has metastasis such as lung, liver metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
3-yr overall survival | 3 years

SECONDARY OUTCOMES:
Disease progression-free survival | 3 years
Local progression-free survival | 3 years
Number and grade of Participants with Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kuai Le Zhao, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen Y, Ye J, Zhu Z, Zhao W, Zhou J, Wu C, Tang H, Fan M, Li L, Lin Q, Xia Y, Li Y, Li J, Jia H, Lu S, Zhang Z, Zhao K. Comparing Paclitaxel Plus Fluorouracil Versus Cisplatin Plus Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Cancer: A Randomized, Multicenter, Phase III Clinical Trial. J Clin Oncol. 2019 Jul 10;37(20):1695-1703. doi: 10.1200/JCO.18.02122. Epub 2019 Mar 28. PMID 30920880
- [Derived] Chen Y, Zhu Z, Zhao W, Li L, Ye J, Wu C, Tang H, Lin Q, Li J, Xia Y, Li Y, Zhou J, Zhao K. A randomized phase 3 trial comparing paclitaxel plus 5-fluorouracil versus cisplatin plus 5-fluorouracil in Chemoradiotherapy for locally advanced esophageal carcinoma-the ESO-shanghai 1 trial protocol. Radiat Oncol. 2018 Feb 27;13(1):33. doi: 10.1186/s13014-018-0979-0. PMID 29482649